CLINICAL TRIAL: NCT04677244
Title: Impact of Echo-endoscopy Biopsy on the Circulating Tumor Cell Level in the Portal System in Pancreatic Adenocarcinoma Management Care
Brief Title: Echo-endoscopy Biopsy Impact on the Circulating Tumor Cell Level
Acronym: EUS-CTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EUS-CTC-IPC 2019-056
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Cancer of Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: prospective monocentric study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Portal vein blood sample (Experimental)
  Interventions: Procedure: Blood sample in portal vein

INTERVENTIONS:
Procedure: Blood sample in portal vein — A 6 ml blood sample will be taken from the portal vein, before and after the echo-endoscopic biopsy of the pancreatic mass. The second sample will be taken after the biopsy if there is no bile drainage, or after bile drainage if indicated. The delay between the end of the biopsy procedure and the puncture will be 5 minutes. A 6 ml peripheral blood sample will also be taken before and after the endoscopic procedure.

SUMMARY:
The aim of this work is to evaluate the impact of endoscopic procedures on the circulating tumoral cells level in order to evaluate the potential effects of an endoscopic procedure in the management of pancreatic tumors.

DETAILED DESCRIPTION:
The study will include 42 evaluable patients suspected of having pancreatic cancer and for whom an echo-endoscopic biopsy (EUS-FNA) and/or biliary drainage is planned.

In these patients, a 6 ml blood sample will be taken from the portal vein before and after the echo-endoscopic biopsy of the pancreatic mass to determine:

* the level of circulating tumor cells (CTC) per milliliter of blood,
* cytological characteristics of CTCs (isolated, clustered, giant, and clustered including other cell types).

A peripheral blood sample will also be taken to evaluate peripheral CTC levels and cytological characteristics before and after biopsy, as well as one month after biopsy.

Patients will be evaluated every 6 months as part of their follow-up to assess the progression of their pathology and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40-85 years old;
* BMI< 30 kg/m2;
* Patients suspected of having pancreatic cancer for whom an ultrasound endoscopic biopsy and/or biliary drainage is planned;
* Affiliation to, or beneficiary of, a social security scheme.

Exclusion Criteria:

* Woman who is pregnant or likely to become pregnant (without effective contraception) or breastfeeding ;
* Person in an emergency situation, person of full age subject to a legal protection measure, or unable to express consent;
* Biliary drainage or attempt at prior biliary drainage outside the center ;
* Preliminary oncological treatment for pancreatic pathology covered by the study;
* Clinical and/or image-visible (CT/MRI) carcinosis ;
* Ascites visible on imaging (CT/MRI) ;
* Impossibility to undergo the medical follow-up of the trial for geographical, social or psychological reasons;
* Contraindications to an endoscopic procedure.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Procedure impact | 5 minutes after procedure
  Rate of patients with a CTC increase > 4 cells/ml in the portal system after the endoscopic procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice CAILLOL, MD, Principal Investigator — Paoli Calmettes Institute
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No